CLINICAL TRIAL: NCT01019616
Title: A Phase Ⅲ Study of Alternative Non-cross-resistant Adjuvant Chemotherapy for Operable Breast Cancer Non-response to Primary Chemotherapy
Brief Title: Alternative Non-cross-resistant Adjuvant Chemotherapy for Operable Breast Cancer Non-response to Primary Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tao OUYANG (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); Peking Union Medical College Hospital (Other); Chinese Academy of Medical Sciences (Other); Peking University First Hospital (Other); Peking University People's Hospital (Other); Beijing Chao Yang Hospital (Other); 307 Hospital of PLA (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D09050703570904
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Primary Breast Cancer
MeSH Terms: interventions — Paclitaxel; Anthracyclines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Experimental)
  Interventions: Drug: paclitaxel/anthracycline
- Control (No Intervention)

INTERVENTIONS:
Drug: paclitaxel/anthracycline — standard chemotherapy regimen(containing paclitaxel or anthracycline) different from primary chemotherapy(containing anthracycline or paclitaxel)
  Other Names: Alternative Non-cross-resistant Adjuvant Chemotherapy
  Arms: Chemotherapy

SUMMARY:
The purpose of this phase Ⅲ, multi-center, prospective, open-label, randomized,controlled study is to determine whether alternative non-cross-resistant adjuvant chemotherapy can increase distant disease free survival(DDFS) in operable patients non-response to primary chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age ≦65 years
* Biopsy proven lymph node positive, estrogen receptor- positive primary breast cancer
* Must have completed a 4-cycle neo-adjuvant chemotherapy with a standard regimen(containing anthracycline or paclitaxel)
* Must have undergone surgery to remove the primary tumor by either a mastectomy or enlarged local excision
* Postoperative residual positive lymph nodes or G1/G2/G3 of Miller & Payne Grading System
* Adequate recovery from recent surgery
* No history of other malignancies
* No currently uncontrolled diseased or active infection
* Not pregnant or breast feeding, and on appropriate birth control if of child-bearing potential
* Adequate cardiovascular function reserve with a myocardial infarction within the past six month
* Adequate hematologic function with:

  1. Absolute neutrophil count (ANC) ≥1500/mm3
  2. Platelets ≥100,000/ mm3
  3. Hemoglobin ≥10 g/dL
* Adequate hepatic and renal function with:

  1. Serum bilirubin ≤1.5×UNL
  2. Alkaline phosphatase and alanine aminotransferase (ALT) ≤2.5 x ULN. (≤5 x ULN is acceptable in the setting of hepatic metastasis)
  3. BUN between 1.7 and 8.3 mmol/L
  4. Cr between 40 and 110 umol/L
* Knowledge of the investigational nature of the study and Ability to give informed consent
* Ability and willingness to comply with study procedures.

Exclusion Criteria:

* Known or suspected distant metastases
* Concurrent malignancy or history of other malignancy
* Uncontrolled diseases(e.g., heart failure, myocardial infarction within 6 months, arrhythmia, unstable diabetes, hypercalcemia) or active infection
* Geographical, social, or psychological problems that would compromise study compliance
* Known or suspected hypersensitivity to anthracycline or paclitaxel

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-03-04 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
distant disease-free survival (DDFS) | 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, Doctor, Study Chair — Beijing Cancer Hospital Breast Center
Locations (7):
- China (7):
  - 307 Hospital of Pla, Beijing
  - Beijing Cancer Hospital Breast Center, Beijing
  - Beijing Chao-Yang Hospital, Beijing
  - Cancer Institution and Hospital.Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People'S Hospital, Beijing